CLINICAL TRIAL: NCT05519657
Title: Incidence and Risk Factors of Postoperative Pulmonary Complications in Elderly Patients Undergoing Robot Assisted Laparoscopic Pelvic Surgery: a Single Center, Prospective, Observational Study
Brief Title: Incidence and Risk Factors of PPCs in Elderly Patients Undergoing Robot Assisted Laparoscopic Pelvic Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Feng Gao, Professor, Tongji Hospital
Other Study IDs: TJ2021S127
Record Dates: First submitted 2021-07-09; First posted 2022-08-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Postoperative Pulmonary Complications; Risk Factors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- postoperative pulmonary complications group: Postoperative pulmonary complications group no intervention
- non-postoperative pulmonary complications group: Non-postoperative pulmonary complications group no intervention

INTERVENTIONS:
Other:
  Groups: non-postoperative pulmonary complications group

SUMMARY:
Postoperative pulmonary complications are important factors affecting the prognosis of patients undergoing surgery. Studies have shown that patients undergoing abdominal or pelvic surgery, emergency surgery, or prolonged surgery are more likely to develop PPCs, especially when robot-assisted laparoscopic surgery is performed at extreme head low. The incidence of PPCs and associated risk factors in patients undergoing robot-assisted laparoscopic surgery compared with those undergoing conventional surgery should be re-examined.

DETAILED DESCRIPTION:
PPCs include bronchospasm, atelectasis, lung infections (bronchitis and pneumonia), exacerbation of pre-existing chronic lung disease, the need for mechanical ventilation after surgery, and respiratory failure. Risk factors for PPCs include preoperative and intraoperative factors. Preoperative was mainly related to the primary status of patients, including age, weight, ASA grade, organ function status, medication history, hypoproteinemia, and concomitant chronic kidney disease, congestive heart failure, COPD, asthma, pulmonary interstitial disease, pulmonary hypertension, and OSA. In this study, elderly patients undergoing robot-assisted laparoscopic pelvic surgery under general anesthesia were selected to prospectively collect basic characteristics, preoperative examination results and perioperative data, and determine the incidence and risk factors of PPCs in this high-risk population cohort. The aim of our study was to determine the incidence of PPCs in elderly patients undergoing robot-assisted laparoscopic pelvic surgery and to screen for associated risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years old
* Selective patients undergoing robot-assisted laparoscopic pelvic surgery under general anesthesia

Exclusion Criteria:

* Patients undergoing oxygen therapy or mechanical ventilation before surgery
* Patients who have received other surgical operations within 30 days
* Patients who have previously undergone lung surgery

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Preoperative: age, sex, height, weight, ASA grade, smoking history, preoperative comorbidities (hypertension, diabetes, coronary heart disease, chronic kidney disease, cerebrovascular disease, COPD), medication history, pulse oxygen saturation, white blood cell count, hemoglobin level, albumin level.
  Intraoperative: operation time (cut skin to sew leather end), anesthesia time (anesthesia induction to tracheal extubation), mechanical ventilation parameters, completion of vital signs, muscle relaxant antagonism, whether the implementation of regional block, infusion, blood loss, amount of urine, perioperative medications (opioids dosage adjustments based on weight and anesthesia time).
Sampling Method: Probability Sample
Enrollment: 154 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of PPCs | Up to 7 days
  One or more of the following conditions occurred: clinically diagnosed PPCs (pneumonia, bronchospasm, ARDS), radiographically diagnosed PPCs (atelectasis, pneumothorax, pleural effusion), postoperative respiratory insufficiency (requiring oxygen or non-invasive mechanical ventilation for more than 1 day), and postoperative tracheal intubation again;Respiratory infections: new or altered sputum properties, new or altered lung shadows, fever, white blood cell >12 × 109/L;Respiratory failure: partial pressure of oxygen in the arterial blood while inhaling air< 60 mmHg, pulse oxygen saturation< 90%, or PaO2/FiO2 < 300;Atelectasis, pneumothorax, pleural effusion: Chest X - ray diagnosis;Bronchospasm: wheezing sound can be relieved with bronchodilators.

SECONDARY OUTCOMES:
Risk factors of PPCs | Up to 7 days
  Risk factors of PPCs in elderly patients undergoing robot assisted laparoscopic pelvic surgery

OTHER OUTCOMES:
Mortality rate within 28 days from the date of surgery | Within 28 days from the date of surgery.
  Within 28 days from the date of surgery, record the number of patients who died due to any cause and total number of observed cases. These two groups of clinical data will be combined to report "mortality rate" in "number of death cases/total number of observed cases".
Mortality rate within 90 days from the date of surgery | Within 90 days from the date of surgery.
  Within 90 days from the date of surgery, record the number of patients who died due to any cause and total number of observed cases. These two groups of clinical data will be combined to report "mortality rate" in "number of death cases/total number of observed cases".

IPD SHARING:
Plan to Share IPD: Undecided